CLINICAL TRIAL: NCT02545374
Title: Medico-economic Evaluation of the DOMOPLAIES Project by the CICAT-LR Network
Brief Title: Medico-economic Evaluation of a Project of Wounds by a Remote Network
Acronym: DOMOPLAIES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 9250
Record Dates: First submitted 2015-09-02; First posted 2015-09-10 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Resident of Languedoc-roussillon; Carrying a Chronic Wound
Keywords: chronic wound; tablet; telemedicine; wounds consultation; Smartphone
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine (Experimental): In the telemedicine arm, all patients will be supported by Telemedicine protocol according to the development of telemedicine in the region.
  The use of teleconsultation allows the couple expert doctor / nurse expert to perform a complex of wound assessment consultation and / or chronic. The use of telemedicine allows for acts of telecare, when the nurse applicant sought a remote support of an expert nurse (under the responsibility of a doctor) for the realization of an act. The use of tele-expertise enables physicians to remotely bring special expertise to improve patient care.
  Interventions: Other: Telemedicine
- Control (Active Comparator): In the control arm, patient care depend on his home, as is currently the case:
  * If it is in the action zone of Cicat-LR network, then it will be supported by an expert nurse of the network that are physically visit the patient's home-lon is the protocols established by the network.
  * If not, then it will be supported by the customs of the attending physician and nursing teams who follow him.
  Interventions: Other: Control

INTERVENTIONS:
Other: Telemedicine
  Arms: Telemedicine
Other: Control
  Arms: Control

SUMMARY:
Estimate in 6 months the impact of the telemedicine on the cure rate of the chronic wounds compared with the usual care(with or without CICAT-LR Network).

ELIGIBILITY:
Inclusion Criteria:

* Being adult
* Taken up residence on the Languedoc-Roussillon
* Patient carrying a wound with healing or improvement objective (wound closure or the appearance of 40% of granulation)
* Informed consent signed,
* Patient member of the Security Social
* Patient having a visiting nurse.

Exclusion Criteria:

* Patient in vital or functional emergency situation during the first call or during the consultation
* Tumoral wound
* dialysis patient
* Arteritis of stage 4 and not revascularizable
* Absence of regular doctor and visiting nurse
* patient refusal
* Refusal of one of the health professionals participating in the pathology care
* Anybody incapable to communicate and to answer the questions
* Pregnant or nursing woman
* Subject deprived of freedom by court or administrative order
* Major subject protected by the law
* For the patients in telemedicine: refusal of the collaboration agreement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Rate of healed chronic wounds during a telemedicine care | Six months after inclusion
  Rate of healed chronic wounds during a telemedicine care versus during a usual medical care
Rate of healed chronic wounds during a usual medical care | Six months after inclusion
  Rate of healed chronic wounds during a telemedicine care versus during a usual medical care

SECONDARY OUTCOMES:
Result to the questionnaire on the quality of life: EQ-5D | Six months after inclusion
  Compare the quality of life of patients with chronic wounds during a telemedicine coverage versus during a usual medical care, thanks to the EQ-5D quality life scale.
A measure of the costs of the management of the disease | Seven months after the inclusion of the last patient
  A measure of the costs of the management of the disease (consumer care, hospitalization, transport ...)
A measure of the costs of the intervention assessed | Seven months after the inclusion of the last patient
  A measure of the costs of the intervention assessed (investment, maintenance, training ...).
The total healing time | Six months after inclusion
The decrease in centimeters of the wound surface to 6 months | Six months after inclusion
The response time between making an appointment and support | Six months after inclusion
The mortality rate within 6 months | Six months after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Wound healing Department, Montpellier, France